CLINICAL TRIAL: NCT07256860
Title: Influence of Chest X-ray vs. Chest CT Scan on the Management of ICU Patients With Respiratory Failure: A Retrospective Study.
Brief Title: Influence of Chest X-ray vs. Chest CT Scan on the Management of ICU Patients With Respiratory Failure
Status: Not yet recruiting | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, sara dichtwald, Dr, Meir Medical Center
Other Study IDs: MMC-0240-25
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Respiratory Failure
Keywords: chest x ray
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Chest computed tomography scan — Performing chest computed tomography scan in addition to chest x-ray in critically ill patients with acute respiratory failure

SUMMARY:
Patients admitted to the intensive care unit (ICU) often require CT imaging. Performing this test on a critically ill patient involves risks, such as those associated with transferring a ventilated and unstable patient (respiratory or hemodynamic instability during transfer, unplanned extubation, unplanned removal of central catheters, drains, etc.), and those associated with intravenous contrast injection (renal impairment, anaphylactic reaction). Additionally, multiple CT scans may create a burden on the radiology department and medical staff, cause CT scans to be postponed for other patients, and increase hospitalization costs (1).

In a study conducted in 2014, approximately 533 CT scans were performed for 359 patients admitted to the ICU at 2 different medical centers. In this study, they examined the extent to which CT scanning affected patient care management by comparing the medical diagnosis given to the patient before and after the scan.

The diagnostic yield of the scan was 40% complete agreement between the diagnosis before and after the CT scan, about 6% partial agreement, and about 54% inconsistency. The CT scan resulted in new findings in the patient's diagnosis in 23% of cases, and in 54% of patients, the CT scan resulted in a change in the patient's treatment plan.

Among the patients who underwent a CT scan, about 23% experienced side effects or adverse events as a result of the scan, of which 6% were defined as life-threatening. The more critically ill the patient was, the greater the risk of these events (1).

In another study, which looked at a subgroup of septic patients in intensive care, there was no agreement between CT findings and the patients' treatment outcomes, and there was no significant effect of the CT scan on the patient's treatment plan (2).

In our previous work on all patients who underwent CT scans in the unit, we found that, in general, the rate of impact of CT scans on the patient's treatment plan was low compared to other studies, although in the group of patients hospitalized due to sepsis, the rate was similar - about a third of the patients. Among the patients hospitalized with multisystem trauma, about 31% of the patients had new traumatic findings on CT scans, but in only half of these patients did the test lead to a change in the treatment plan. It appears from this work that the group in which it was possible to retrospectively find the largest number of CT scans that could have been omitted was the group of patients with respiratory failure. The purpose of performing CT scans in these patients was mainly to look for pulmonary infiltrates, pleural effusions, or pulmonary embolism. With the exception of pulmonary embolism, a condition that is relatively rare compared to other diagnoses in patients with acute respiratory failure, the other diagnoses could also be confirmed by physical examination, ultrasound examination, or chest x-ray (these patients usually undergo a chest x-ray as part of the investigation of acute respiratory failure anyway), and this may be the reason why the CT scan did not add relevant information to change the treatment plan in these patients. However, we did not specifically examine in this study whether the chest x-ray showed all the findings seen on the chest CT scan, and whether the CT scan added new findings, and especially whether these new findings would have changed the treatment plan (such as pulmonary embolism). In this study, we would like to focus on this group of patients.

ELIGIBILITY:
Inclusion Criteria: All patients who underwent CT scans as part of their hospitalization in the intensive care unit for acute respiratory failure/hypoxemia, from January 2020 to January 2023.

-

Exclusion Criteria: Missing data.

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients who underwent CT scans as part of their hospitalization in the intensive care unit for acute respiratory failure/hypoxemia, from January 2020 to January 2023.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-11-21 (Estimated); Primary Completion 2026-11-25 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
New findings in chest CT scan vs. chest x-ray | 1 year
  To examine, among intensive care patients who underwent a chest CT scan for the purpose of investigating respiratory failure/hypoxemia, whether the CT scan revealed new findings that were not seen on a chest x-ray performed immediately prior to the scan, and whether these findings changed the patient's treatment.
New findings in chest CT scan vs. chest x-ray and implications on therapy | 1 year
  To examine, among intensive care patients who underwent a chest CT scan for the purpose of investigating respiratory failure/hypoxemia, whether the CT scan revealed new findings that were not seen on a chest x-ray performed immediately prior to the scan, and whether these findings changed the patient's treatment.